CLINICAL TRIAL: NCT00538499
Title: Optimal Pain Management After Video-Assisted Thoracic Surgery
Brief Title: Fentanyl With or Without Bupivacaine in Reducing Pain in Patients Undergoing Video-Assisted Chest Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000565803; RPCI-I-37404
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Pain; Perioperative/Postoperative Complications
Keywords: pain; perioperative/postoperative complications
MeSH Terms: conditions — Pain; Postoperative Complications | interventions — Fentanyl; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fentanyl citrate (Other)
  Interventions: Drug: Fentanyl citrate
- bupivcaine hydrochloride (Experimental)
  Interventions: Drug: Bupivacaine hydrocloride
- videothoracoscopy (Other)
  Interventions: Procedure: videothoracoscopy

INTERVENTIONS:
Drug: Fentanyl citrate
  Arms: Fentanyl citrate
Drug: Bupivacaine hydrocloride
  Arms: bupivcaine hydrochloride
Procedure: videothoracoscopy
  Arms: videothoracoscopy

SUMMARY:
RATIONALE: Patient-controlled analgesia using fentanyl and bupivacaine may lessen pain caused by video-assisted chest surgery. Giving bupivacaine in different ways may give better pain relief.

PURPOSE: Thisrandomized clinical trial is comparing three different ways to give bupivacaine together with fentanyl to see how well they work in reducing pain after video-assisted chest surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the efficacy of intravenous, patient-controlled, narcotic pain management alone to the efficacy of intermittent bolus injection of bupivacaine hydrochloride via an intrapleural catheter in patients who have successfully undergone video-assisted thoracic surgery (VATS).

Secondary

* To compare the efficacy of intermittent bolus administration of bupivacaine hydrochloride to the efficacy of continuous bupivacaine hydrochloride administration via an intrapleural catheter in patients who have successfully undergone VATS.
* To compare visual analog scale pain scores at all measurement times.
* To compare patient satisfaction scores for each method of pain control.
* To compare rates of conversion from bolus delivery to intravenous narcotic delivery.
* To compare rates of conversion from continuous intrapleural infusion to bolus delivery or intravenous narcotic delivery alone.
* To compare the total amount of narcotics used between bolus intrapleural delivery and continuous intrapleural infusion.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive intravenous patient-controlled analgesia (IV-PCA) fentanyl citrate beginning once the patient is awake and alert after surgery and continuing for 24 hours.
* Arm II: Patients receive intermittent intrapleural bolus bupivacaine hydrochloride immediately after surgery and then at 6, 12, 18, and 24 hours after surgery and IV-PCA fentanyl citrate as in arm I.
* Arm III: Patients receive a continuous infusion of intrapleural bupivacaine hydrochloride beginning immediately after surgery and continuing for 24 hours and IV-PCA fentanyl citrate as in arm I.

In all arms, visual analog scale measurements are taken at baseline and 6, 12, 18, and 24 hours post-surgery. After 24 hours, a 5-point Likert scale survey is administered to assess overall patient satisfaction with pain control in the 24-hour postoperative period.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Candidate for video-assisted thoracic surgery (VATS) and unlikely to require conversion to open thoracotomy as determined by physician
* Able to satisfactorily complete a Visual Analog Scale (VAS) measurement

  * Patients who are too sedated postoperatively or who are unable to properly mark a VAS scale due to other factors (poor eyesight, lack of manual dexterity, or lack of comprehension of the test) are ineligible

PATIENT CHARACTERISTICS:

* No allergy to bupivacaine hydrochloride or fentanyl citrate
* No known renal or liver disease (i.e., hepatic insufficiency or cirrhosis) that would affect metabolism of drugs used in this study
* Not pregnant or nursing
* Negative pregnancy test
* No thoracic infection within the past 3 months
* Weight ≥ 55 kg
* ALT and AST < 10% of upper limit of normal
* Serum creatinine < 1.5 mg/dL
* BUN < 40 mg/dL

PRIOR CONCURRENT THERAPY:

* No concurrent narcotics for pain management
* No concurrent amiodarone, barbiturate anesthetics or other CNS depressants, diazepam, droperidol, nitrous oxide, or protease inhibitors

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10-28 (Actual); Primary Completion 2007-07-27 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Overall consumption of narcotics between the 3 treatment arms | up to 24 hours after surgery

SECONDARY OUTCOMES:
Differences in Visual Analog Scale measurements between the 3 treatment arms | baseline and 6, 12, 18, and 24 hours post-surgery
Rates of conversion and overall satisfaction with pain management | 24 hours post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Todd L. Demmy, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States